CLINICAL TRIAL: NCT03446196
Title: Hemodynamic Optimization During Single Kidney Transplantation With MostcareUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Medical Doctor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4423/AO/18
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Transplant Dysfunction
Keywords: Transplantation, Fluid Balance

STUDY DESIGN:
Intervention Model Description: Adult patients with end stage kidney disease undergoing single kidney transplantation from deceased donor. Two arms. One arm will undergo fluid replacement based on mostcare UP information, other arm will undergo fluid replacement based on clinician experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MOSTCARE UP (Experimental): Clinician will be able to read MOSTCARE parameters and to choose the best treatment to adequate hemodynamics considering that current literature suggests a fluid IV expansion only if PPV > 12%
  Interventions: Device: Fluid replacement based on MOSTCARE up
- CLINICIAN EXPERIENCE (No Intervention): Fluid replacement will be made based on clinician experience

INTERVENTIONS:
Device: Fluid replacement based on MOSTCARE up — Clinician will be able to read MOSTCARE parameters and to choose the best treatment to adequate hemodynamics considering that current literature suggests a fluid IV expansion only if PPV > 12%
  Arms: MOSTCARE UP

SUMMARY:
There are currently no clear recommendations on hemodynamic targets during kidney transplantation and most anesthesiologists rely on empiric or obsolete parameters such as CVP.

The aim of this study is to investigate hemodynamic management of these patients applying a new generation of advanced monitoring systems such as MOSTCAREUP which can potentially provide a clear overview of the circulatory status beat by beat and to adjust fluid therapy in every single patient or clinical condition.

DETAILED DESCRIPTION:
Renal transplantation is actually considered the optimal elective treatment for end stage kidney disease.

Successful renal transplantation involves the optimization of several parameters. Previous studies have suggested that perioperative hemodynamic factors influence immediate and long-term graft survival.

Perioperative hemodynamic management of this kind of surgery is nowadays focused on optimization of fluid therapy concerning both the donor and the graft and their interaction. Postoperative graft function is not exclusively determined by donor and graft characteristics. Several studies over the last 30 years indeed demonstrated that hemodynamic status of the recipient during kidney transplant surgery relates to graft function and proper management of balancing fluid plays a critical role through maintaining optimal blood volume and so assure an adequate supply of oxygen to the tissues.

Aggressive expansion of the intravascular volume during transplantation surgery has been recommended by most previous studies supporting the so called "liberal" approach to fluid management suggesting that a massive intravascular volume expansion was necessary improve renal blood flow and minimize hypoperfusion caused tissue damages. Nowadays it is clear that adequate early graft function requires perfusion of the transplanted kidney, which may be enhanced by expansion of the intravascular volume in the recipient. However, some studies have reported that aggressive intraoperative volume expansion is not always warranted in kidney transplantation and can expose patients with preexistent cardiac disease or poor myocardial function to the risk of fluid overload, acute respiratory failure, and prolonged ventilation. Moreover fluid overload has been demonstrated to be harmful even for graft perfusion, microcirculation and tissue oxygen delivery.

There are currently no clear recommendations on hemodynamic targets during kidney transplantation and most anesthesiologists rely on empiric or obsolete parameters such as CVP.

The aim of this study is to investigate hemodynamic management of these patients applying a new generation of advanced monitoring systems such as MOSTCAREUP which can potentially provide a clear overview of the circulatory status beat by beat and to adjust fluid therapy in every single patient or clinical condition.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent Renal transplantation candidate

Exclusion Criteria:

Double kidney transplantation Living donor kidney transplantation Hystory of heart failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Urine output in the first hour post unclamping (ml) in the two groups | first hour post unclamping during kydney transplanation
  Urine output in the first hour post unclamping (ml) in the two groups

SECONDARY OUTCOMES:
1) Urine output in the first 24h (ml) | 24hour
  1) Urine output in the first 24h (ml)
2) Need for haemodialysis in the first week (% of patients) | 7 days
  2) Need for haemodialysis in the first week (% of patients)
3) First week creatinine and urea trend in the two groups | 7 days
  3) First week creatinine and urea trend in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Padua, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Undecided
All datas will be probably shared at the end of the study

REFERENCES:
- [Background] Calixto Fernandes MH, Schricker T, Magder S, Hatzakorzian R. Perioperative fluid management in kidney transplantation: a black box. Crit Care. 2018 Jan 25;22(1):14. doi: 10.1186/s13054-017-1928-2. PMID 29368625
- [Background] Schnuelle P, Johannes van der Woude F. Perioperative fluid management in renal transplantation: a narrative review of the literature. Transpl Int. 2006 Dec;19(12):947-59. doi: 10.1111/j.1432-2277.2006.00356.x. PMID 17081224
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972

DOCUMENTS (1):
  • Study Protocol (2018-02-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03446196/Prot_001.pdf